CLINICAL TRIAL: NCT05021835
Title: ZEUS - Effects of Ziltivekimab Versus Placebo on Cardiovascular Outcomes in Participants With Established Atherosclerotic Cardiovascular Disease, Chronic Kidney Disease and Systemic Inflammation
Brief Title: ZEUS - A Research Study to Look at How Ziltivekimab Works Compared to Placebo in People With Cardiovascular Disease, Chronic Kidney Disease and Inflammation
Acronym: ZEUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX6018-4758; U1111-1259-3422 (Other: World Health Organization (WHO)); 2023-506926-35 (Other: European Medical Agency (EMA)); jRCT2021210033 (Registry Identifier: JAPIC)
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Risk; Chronic Kidney Disease; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ziltivekimab (Experimental): Participants will receive Ziltivekimab B or Ziltivekimab C subcutaneously once monthly for up to 4 years.
  Interventions: Drug: Ziltivekimab B; Drug: Ziltivekimab C
- Placebo (Placebo Comparator): Participants will receive either placebo (Ziltivekimab B) or placebo (Ziltivekimab C) subcutaneously once monthly for up to 4 years.
  Interventions: Drug: Placebo (Ziltivekimab B); Drug: Placebo (Ziltivekimab C)

INTERVENTIONS:
Drug: Ziltivekimab B — Administered subcutaneously (s.c., under skin) once-monthly added to standard of care.
  Arms: Ziltivekimab
Drug: Ziltivekimab C — Administered subcutaneously (s.c., under skin) once-monthly added to standard of care.
  Arms: Ziltivekimab
Drug: Placebo (Ziltivekimab B) — Administered subcutaneously (s.c., under skin) once-monthly added to standard of care.
  Arms: Placebo
Drug: Placebo (Ziltivekimab C) — Administered subcutaneously (s.c., under skin) once-monthly added to standard of care.
  Arms: Placebo

SUMMARY:
This study is conducted to see if ziltivekimab reduces the risk of having cardiovascular events (for example heart attack and stroke) in people with cardiovascular disease, chronic kidney disease and inflammation.

Participants will either get ziltivekimab (active medicine) or placebo (a dummy medicine which has no effect on the body). This is known as the study medicine. Which treatment participants get is decided by chance. Participants chance of getting ziltivekimab or placebo is the same.

Ziltivekimab is not yet approved in any country or region in the world. It is a new medicine doctors cannot prescribe.

Participants will get the study medicine in a pre filled syringe. Participants will need to use the pre filled syringe to inject the study medicine into a skinfold once-monthly.

The study is expected to last for up to 4 years. Participants will have up to 20 clinic visits. Participants will have blood and urine samples taken at most of the clinic visits.

Participants will have their heart examined using sound waves (echocardiography) and electrodes (electrocardiogram).

Women cannot take part if pregnant, breast-feeding or planning to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease defined by one of the below:

  1. Estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 15 and below 60 mL/min/1.73 m^2 (using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation)
  2. Urinary albumin-to-creatinine ratio (UACR) >= 200 milligrams per gram (mg/g) and eGFR >= 60 mL/min/1.73 m2 (using the CKD-EPI creatinine equation)
* Serum high-sensitivity C-reactive protein (hs-CRP) greater than or equal to 2 milligram per liter (mg/L)
* Evidence of atherosclerotic cardiovascular disease (ASCVD) by one or more of the following:

  a) Coronary heart disease defined as at least one of the following: i. Documented history of MI ii. Prior coronary revascularisation procedure iii. greater than or equal to 50% stenosis in major epicardial coronary artery documented by cardiac catheterisation or CT coronary angiography b) Cerebrovascular disease defined as at least one of the following: i. Prior stroke of atherosclerotic origin ii. Prior carotid artery revascularisation procedure iii. greater than or equal to 50% stenosis in carotid artery documented by X-ray angiography, MR angiography, CT angiography or Doppler ultrasound.

  c) Symptomatic peripheral artery disease (PAD) defined as at least one of the following: i. Intermittent claudication with an ankle-brachial index (ABI) below or equal to 0.90 at rest ii. Intermittent claudication with a greater than or equal to 50% stenosis in peripheral artery (excluding carotid) documented by X-ray angiography, MR angiography, CT angiography or Doppler ultrasound iii. Prior peripheral artery (excluding carotid) revascularisation procedure iv. Lower extremity amputation at or above ankle due to atherosclerotic disease (excluding e.g. trauma or osteomyelitis).

Exclusion Criteria:

* Clinical evidence of, or suspicion of, active infection at the discretion of the investigator.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris, or transient ischaemic attack within 60 days prior to randomisation (visit 2).
* Planned coronary, carotid or peripheral artery revascularisation known on the day of randomisation (visit 2).
* Major cardiac surgical, non-cardiac surgical, or major endoscopic procedure (thoracoscopic or laparoscopic) within the past 60 days prior to randomisation (visit 2) or any major surgical procedure planned at the time of randomisation (visit 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6200 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of 3-point Major Adverse Cardiovascular Event (MACE), a composite endpoint consisting of: Cardiovascular (CV) death, non-fatal Myocardial Infarction (MI) and non-fatal stroke | From randomisation (month 0) to end-of-study (up to 48 months)
  Months

SECONDARY OUTCOMES:
Time to first occurrence of expanded MACE, a composite endpoint consisting of: CV death, non-fatal MI, non-fatal stroke and hospitalisation for unstable angina pectoris requiring urgent coronary revascularisation | From randomisation (month 0) to end-of-study (up to 48 months)
  Months
Number of heart failure hospitalisations or urgent heart failure visits or CV deaths | From randomisation (month 0) to end-of-study (up to 48 months)
  Count
Time to first occurrence of a composite kidney endpoint consisting of: CV death, onset of persistent atleast 40 percent (%) reduction in eGFR (CKD-epidemiology collaboration [CKD-EPI]) compared with baseline, kidney failure | From randomisation (month 0) to end-of-study (up to 48 months)
  Months
Time to occurrence of all-cause mortality | From randomisation (month 0) to end-of-study (up to 48 months)
  Months
Time to first occurrence of each of the individual components of the expanded MACE endpoint and the kidney composite endpoint. | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Time to first occurrence of MI (fatal and non-fatal). | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Time to first occurrence of stroke (fatal and non-fatal). | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Time to first occurrence of a composite MACE endpoint consisting of: all-cause mortality, non-fatal MI and non-fatal stroke | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Time to first occurrence of a 4-component kidney endpoint consisting of: onset of persistent at least 40% reduction in eGFR (CKD-EPI) compared with baseline, kidney failure | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Time to first occurrence of coronary revascularisation | From randomisation (month 0) to end-of-study (up to 48 months).
  Months
Change in Urinary Abumin-to-Ceatinine ratio (UACR). | From randomisation (month 0) to 2 years (24 months).
  Percentage
Change in eGFR (CKD-EPI)) | From randomisation (month 0) to 2 years (24 months)
  mL/min/1.73 m^2
Annual rate of change in eGFR (CKD-EPI) (total eGFR slope) | From randomisation (month 0) to end-of-study (up to 48 months).
  mL/min/1.73 m^2/ year
Change in high-sensitivity C-reactive protein (hs-CRP) | From randomisation (month 0) to 2 years (24 months
  Percentage
Change in N-terminal-pro-brain natriuretic peptide ( NT-pro-BNP) | From randomisation (month 0) to 2 years (24 months)
  Percentage
Change in left ventricular ejection fraction (LVEF) | From randomisation (month 0) to 2 years (24 months)
  Percentage
Number of events of atrial fibrillation | From randomisation (month 0) to end-of-study (up to 48 months).
  Count
Change in haemoglobin | From randomisation (month 0) to 2 years (24 months)
  Grams per deciliter (g/dL)
Number of hospitalisations with infection as primary cause or death due to infection. | From randomisation (month 0) to end-of-study (up to 48 months).
  Count
Change in Short Form 36 (SF-36) Physical Component Score (PCS) | From randomisation (month 0) to 2 years (24 months)
  Score on scale

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1019):
- United States (180):
  - Uni of Alabama at Birmingham, Birmingham, Alabama
  - Chambliss Clinical Trials, LLC, Montgomery, Alabama
  - Lenzmeier Fam Med CCT Research, Glendale, Arizona
  - Aventiv Research Inc., Mesa, Arizona
  - Univ of Arkansas Med Sciences, Little Rock, Arkansas
  - Unity Health-Searcy Medical Center, Searcy, Arkansas
  - National Heart Institute Cal, Beverly Hills, California
  - California Inst Of Renal Res, Chula Vista, California
  - California Institute of Renal Research #10, Chula Vista, California
  - Valley Clinical Trials, Covina, California
  - Valiance Clinical Research, Huntington Park, California
  - Scripps Wht Diab Inst La Jolla, La Jolla, California
  - Balboa Nephro Med Gr Inc LaMes, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - VA Loma Linda Hlthcr Sys, Loma Linda, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Angel City Research, Inc., Los Angeles, California
  - North America Research Institute, Lynwood, California
  - Hoag Medical Group, Newport Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Riverside Nephrology Physicians, Riverside, California
  - N America Res Inst - San Dimas, San Dimas, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - Denver Health Outpatient Medical Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - VA-Connecticut (VACHS), West Haven, Connecticut
  - George Washington Uni Med, Washington D.C., District of Columbia
  - Excel Med Ctr Clinical Trials, Boca Raton, Florida
  - Innovative Research of W FL, Clearwater, Florida
  - Florida Premier Cardiology, Delray Beach, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Integrative Research Assoc Inc, Fort Lauderdale, Florida
  - Elixia Pines, Hollywood, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - Northeast Research Institute, Jacksonville, Florida
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - Clinical Research of Cent FL, Lakeland, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Life Spring Research, Miami, Florida
  - Allied Biomedical Research, Miami, Florida
  - San Marcus Res Clin Miami Lakes, Miami Lakes, Florida
  - Office of Kenneth Blaze DO, Miramar, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - A&R Research Group, LLC, Pembroke Pines, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - East Coast Institute for Research LLC_St. Augustine, Saint Augustine, Florida
  - St Johns Center for Clin. Res, Saint Augustine, Florida
  - Javara/Privia Med Grp GA,LLC, Albany, Georgia
  - Southeastern Clinical R.I., Augusta, Georgia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Hope Clin Res & Wellness, Conyers, Georgia
  - Javara Inc._Albany, Fayetteville, Georgia
  - NSC Research, Inc, Johns Creek, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - Javara Inc._Winston Salem, Savannah, Georgia
  - Saltzer Medical Group Research, Nampa, Idaho
  - Endeavor Health Clinical Operations-NCH, Arlington Heights, Illinois
  - Research by Design LLC, Chicago, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Endeavor Health, Skokie, Illinois
  - Central Illinois Diabetes and Clinical Research, Springfield, Illinois
  - Clin Invest Spec, Inc, Wauconda, Illinois
  - MediSphere Medical RC, Evansville, Indiana
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - Midwest Heart & Vasc Spec, Overland Park, Kansas
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - Lexington VA Health Care System, Lexington, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Norton Heart Specialists-Springs, Louisville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Clinical Trials of Ame, LLC, Monroe, Louisiana
  - IMA Clinical Research, Monroe, Louisiana
  - Grace Research, LLC_Shreveport, Shreveport, Louisiana
  - Louisiana Heart Center_Slidell, Slidell, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - John P Hakim MD and Associates, Clinton, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Henry Ford Hospital_Detroit, Detroit, Michigan
  - Elite Research Center, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - McLaren Northern MI Hosp, Petoskey, Michigan
  - AHS dba Abbot NW Hosp Diab Cen, Minneapolis, Minnesota
  - University of Minnesota_Minneapolis_1, Minneapolis, Minnesota
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Gateway CV Research Cntr Inc., St Louis, Missouri
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - Nebraska Heart Institute_Lincoln, Lincoln, Nebraska
  - VA NEB - Western IA Health Stm, Omaha, Nebraska
  - Methodist Phys Clin Heart Cons, Omaha, Nebraska
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Uni of New Mexico-Clinical, Albuquerque, New Mexico
  - NYU Nephrology Associates, Mineola, New York
  - NYU Grossman School of Med, New York, New York
  - Mount Sinai Hosp at NYC, New York, New York
  - Northport VA Med Ctr Northport, Northport, New York
  - Mattoo & Bhat M.A., Ridgewood, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - DaVita Clinical Research - New York, The Bronx, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - Kernodle Clin Dpt-Pvt Diagnost, Burlington, North Carolina
  - UNC- Chapel Hill, Chapel Hill, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Javara Inc._Charlotte, Charlotte, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Univ of Cincinnati Med Cent, Cincinnati, Ohio
  - VA Northeast Ohio Healthcare System (VANEOHS), Cleveland, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Aria Endocrine Metabolic Assoc, Philadelphia, Pennsylvania
  - Parkside Family Medicine, Philadelphia, Pennsylvania
  - Ocean St Clin Res Partnrs, LLC, Lincoln, Rhode Island
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - Palmetto Clinical Research, Greenville, South Carolina
  - Family Medicine of SayeBrook LLC, Myrtle Beach, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Balad Hlth Sys-Welmont CardCVA, Greeneville, Tennessee
  - Tennova HC Turkey Creek MC, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - CV Research of Knoxville, Powell, Tennessee
  - Liberty Research Center, Arlington, Texas
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Novel Research LLC, Bellaire, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Research Trials Worldwide LLC, Cypress, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - Thyroid Endocrinology & Diabetes PA, Dallas, Texas
  - Liberty Research Center_Dallas, Dallas, Texas
  - DHR Health Inst for Res & Dev, Edinburg, Texas
  - Academy of Diabetes, T&E, El Paso, Texas
  - Care United Research, LLC, Forney, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - Javara /TX.Hlth LLC dba Prvia, Fort Worth, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Baylor College Of Medicine_Houston, Houston, Texas
  - Biopharma Informatic_Houston, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Prolato Clinical Research Cntr, Houston, Texas
  - Card Specialists of Willowbrook, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Biopharma Informatic_Houston_0, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Texas Inst, Kdny & Endo Disor, Lufkin, Texas
  - RGV Endocrine Center, McAllen, Texas
  - Carlos Arauz-Pacheco Md, Pa, Rockwall, Texas
  - Texas Diabetes Institute, San Antonio, Texas
  - Clinical Advancement Ctr, PLLC, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Javara Privia Grp Gulf Cst LLC, San Marcos, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Javara Inc/Privia Md GpLLC Fst, Forest, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Providence Medical Research Center, Spokane, Washington
  - Aspirus Research Institute, Wausau, Wisconsin
  - Marshfield Clinic, Weston, Wisconsin
- Argentina (16):
  - Mautalen Salud e investigación, CABA, Buenos Aires
  - Sanatorio Finochietto, CABA, Buenos Aires
  - Instituto Cardiovascular Buenos Aires, CABA, Buenos Aires
  - CEMEDIC, CABA, Buenos Aires
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Centro de Investigaciones Médicas Clínica de Fracturas y Or, Mar del Plata, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro Medico Lebensohn, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - Centro Médico Viamonte SRL, CABA
  - Centro de Educación Médica e Investigaciones Clínicas Saaved, Capital Federal
  - Cardiología Palermo Duplicate, Ciudad Autónoma de Buenos Aire
  - Instituto Médico DAMIC, Córdoba
  - Instituto Médico CER, Quilmes - Buenos Aires
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán.
  - Instituto de Investigaciones Clinicas San Nicolás, San Nicolás
- Australia (19):
  - The Canberra Hospital_Garran, Garran, Australian Capital Territory
  - Gosford Renal Research, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Applied Research Centre, Westmead, New South Wales
  - Illawarra Heart Health Centre, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Core Research Centre, Milton, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital Cardiovascular Clinical Trials, Adelaide, South Australia
  - HeartCare SA, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health Heart, Clayton, Victoria
  - St Vincent's Hospital_Fitzroy_0, Fitzroy, Victoria
  - Geelong Cardiology Research Unit, Geelong, Victoria
  - Melbourne Renal Research Group, Reservoir, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - La Trobe Regional Hospital, Traralagon, Victoria
  - HeartCare WA (Joondalup), Joondalup, Western Australia
- Belgium (11):
  - AZORG Aalst - Moorselbaan, Aalst
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - AZ Klina - Brasschaat - Cardiology, Brasschaat
  - AZ Sint-Jan - Campus Brugge_Brugge, Bruges
  - AZ Sint-Jan - Campus Brugge, Bruges
  - Ziekenhuis Oost Limburg - Cardiology, Genk
  - Ziekenhuis Oost-Limburg AV - Cardiology, Genk
  - AZ Groeninge - Kortrijk - Cardiology, Kortrijk
  - CHR de la Citadelle, Liège
  - AZ Sint-Maarten Mechelen - Cardiology, Mechelen
  - AZ OOSTENDE (Campus DAMIAAN), Ostend
- Brazil (20):
  - Centro de Diag. e Pesquisa da Osteoporose do Espírito Santo, Vitória, Espírito Santo
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Eurolatino Medical Research Center, Uberlândia, Minas Gerais
  - Instituto Pró-Renal Brasil, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - PUCCAMP - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - Impar Serviços Hospitalares S/A, São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre/ RS
  - HBA S/A Assistência Médica e Hospitalar, Salvador
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo Do Campo/SP
  - Centro de Diabetes e Obesidade - HRim e Hipertensao, São Paulo - SP
- Bulgaria (26):
  - Medical Centre Diamedical-2013, Dimitrovgrad
  - 'Medical center Medi city 21' OOD, Kyustendil
  - Medical center Medi City 21 OOD, Kyustendil
  - "Medical Center Hera" EOOD - Montana, Montana
  - SHATC Sveti Georgi - Pernik OOD, Pernik
  - "Medical center Medconsult Pleven" OOD, Pleven
  - Medical center Medconsult Pleven OOD, Pleven
  - MHAT Heart and Brain, Pleven
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Cardiology, Plovdiv
  - 'MHAT Hadzhi Dimitar' OOD, Sliven
  - MHAT Hadzhi Dimitar OOD, Sliven
  - Mhat "Nch", Sofia
  - "Acibadem City Clinic UMHAT" EOOD, Sofia, Cardiology clinic, Sofia
  - Acibadem City Clinic UMHAT EOOD, Sofia
  - DCC Aleksandrovska EOOD, Sofia
  - UMHAT "Sveti Ivan Rilski" EAD, Sofia
  - UMHAT "Sveti Ivan Rilski", Sofia
  - "Medical Center Hera" EOOD - Sofia, Sofia
  - Medical center ISUL - Tsaritsa Yoanna EOOD, Sofia
  - "UMHAT "Sveta Anna" Sofia" AD, Clinic of Cardiology, Sofia
  - "UMHAT "Sveta Anna" Sofia", Sofia
  - Prevencia - 2000 - MCOC OOD, Stara Zagora
  - Medical Center "Nov Rehabilitatsionen center" EOOD, Stara Zagora
  - Medical Center Nov Rehabilitatsionen center EOOD, Stara Zagora
  - UMHAT "Sveta Marina" EAD, Varna
  - Medical center Berbatov, Yambol
- Canada (30):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Synergy Wellness Clinic, Sherwood Park, Alberta
  - BC Diabetes Canada, Vancouver, British Columbia
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - LMC Diabetes & Endocrinology (Barrie), Barrie, Ontario
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - LMC Clin Res Inc. Thornhill, Concord, Ontario
  - Centricity Research Etobicoke, Etobicoke, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - One Heart Care, Mississauga, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - Partnrs Adv Cardio Eval (PACE), Newmarket, Ontario
  - North York Diagn & Cardiac Ctr, North York, Ontario
  - Oakville Cardiovascular Research LP, Oakville, Ontario
  - LMC Clinical Research Inc. Oakville, Oakville, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Heart Health Institute Research, Inc., Scarborough Village, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
  - Viacar Recherche Clinique Inc., Brossard, Quebec
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Viacar Recherche Clinique Inc., Longueuil, Quebec
  - Centre de recherché du CHUS, Sherbrooke, Quebec
  - Centre de santé et de services, Terrebonne, Quebec
  - Recherche Clinique Sigma inc, Québec
  - Institut universitaire de cardiologie, Québec
  - CHU de Quebec-Universite Laval, Québec
- China (80):
  - Fu Yang People's Hospital-Nephrology, Fuyang, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital-Cardiology, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University-Cardiology, Beijing, Beijing Municipality
  - Peking University Third Hospital-Cardiology, Beijing, Beijing Municipality
  - Beijing Hospital-Nephrology, Beijing, Beijing Municipality
  - Chinses People's Liberation Army General Hospital-Nephrology, Beijing, Beijing Municipality
  - Chinses PLA General Hospital-Nephrology, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University-Cardiology, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University-Nephrology, Xiamen, Fujian
  - Lanzhou University Second Hospital_Internal Medicine-Cardiovascular Dept, Lanzhou, Gansu
  - The Second Hospital & Clinical Medical School, Lanzhou University-Internal Medicine & Cardiovascular, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University-Cardiology, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College-Nephrology, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region-Nephrology Department, Nanning, Guangxi
  - Huizhou Central People's Hospital_Internal Medicine-Cardiovascular Dept, Huizhou, Hainan
  - Xingtai People's Hospital-Nephrology, Xingtai, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology-Nephrology, Luoyang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University-Cardiology, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital-Cardiology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST-Cardiology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST-Nephrology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University-Cardiology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changde City -Internal Medicine-Cardiovascular, Changde, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second People's Hospital of Huai'an-Nephrology, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The People's Hospital of Guangxi Zhuang Autonomous Region-Cardiology Department, Nanning, Jiangsu
  - The First Affiliated Hospital of Soochow University-Cardiology, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University-Cardiology, Xuzhou, Jiangsu
  - The Affiliated Hospital Of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Nephrology, Zhenjiang, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincial People's Hospital-Cardiology, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University-Nephrology, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University-Cardiology, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University-Nephrology, Changchun, Jilin
  - The Second Hospital of Jilin University_Changchun, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University-Nephrology, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Central Hospital of Dalian University of Technology (Dalian Municipal Central Hospital) -Cardiology, Dalian, Liaoning
  - Central Hospital of Dalian University of Technology (Dalian Municipal Central Hospital) -Nephrology, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University-Cardiology, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University-Cardiology, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an JiaoTong University-Cardiovascular, Xi'an, Shaanxi
  - Jinan Central Hospital-Cardiovascular, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital)-Cardiology, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital-Cardiology, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University-Nephrology, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University-Nephrology, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai-Nephrology, Shanghai, Shanghai Municipality
  - Linfen Central Hospital-Cardiology, Linfen, Shanxi
  - Sichuan Provincial People's Hospital- Nephrology, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin 4th Center Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine-Cardiology, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital-Cardiology Department, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Xuanwu Hospital Capital Medical University-Cardiology, Beijing
  - The First People's Hospital of Changde City -Internal Medicine-Cardiovascular, Changde
  - Sichuan Provincial People's Hospital- Nephrology, Chengdu
  - The First Affiliated Hospital, Zhejiang University School of Medicine-Cardiology, Hangzhou
  - Huizhou Central People's Hospital_Internal Medicine-Cardiovascular Dept, Huizhou
  - Jinan Central Hospital Affiliated to Shandong University (Cardiovascular Dept), Jinan
  - The Second Hospital of Shandong University, Jinan
  - The Second Affiliated Hospital of Shantou University Medical College-Nephrology, Shantou
  - Shengjing Hospital of China Medical University, Shenyang
- Croatia (8):
  - KB Dubrava, Zavod za bolesti srca i krvnih zila, Zagreb, City of Zagreb
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Specijalna bolnica Krapinske Toplice - Kardiologija, Krapinske Toplice, Krapinsko Zagorska County
  - KBC Rijeka, Zavod za kardiomiopatije, Rijeka
  - KBC Rijeka, Zavod za nefrologiju, Rijeka
  - KBC Split / Krizine/ Kardiologija, Split
  - KBC Zagreb, Klinika za bolesti srca i krvnih zila, Zagreb
  - KBC Zagreb, Zavod za nefrologiju, Zagreb
- Czechia (6):
  - Edumed Broumov, Broumov
  - KARDIOLOGIE - LIBEREC s.r.o., Liberec
  - EDUMED s.r.o., Náchod
  - IKEM Klinika nefrologie, Prague
  - Medicon a.s., Prague
  - Nemocnice Slany Kardiologie, Slaný
- Denmark (9):
  - Holbæk Sygehus, Holbæk, Region Sjælland
  - Aalborg Universitetshospital Kardiologisk Afdeling, Aalborg
  - Aarhus Universitetshospital, Hjertesygdomme, Aarhus N
  - Regionshospitalet Gødstrup, Hjertesygdomme, Herning
  - Hvidovre Hospital Hjertemedicinsk, Hvidovre
  - Kolding Sygehus Karkirurgi, Kolding
  - Sjællands Universitetshospital_Roskilde, Roskilde
  - Kardiologisk Odense & Svendborg, Svendborg
  - Viborg Sygehus, Viborg
- Germany (36):
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau, Baden-Wurttemberg
  - SRH Klinikum Karlsbad-Langensteinbach GmbH - Innere Medizin, Karlsbad, Baden-Wurttemberg
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein, Holstein
  - Sana Kliniken Oberfranken Coburg GmbH - II. Med. Klinik, Kardiologie, Coburg, Thuringia
  - Uniklinik Aachen - Med. Klinik I, Aachen
  - Universitaetsklinikum Aachen AöR, Aachen
  - Kardiologische Praxis, Bad Homburg, Bad Homburg
  - Charité - Campus Benjamin Franklin - Klinik für Nephrologie und Internistische Intensivmedizin, Berlin
  - Praxis Dr.med. Frank Menzel, Dessau
  - Facharztzentrum Dresden Betriebsgesellschaft mbH, Dresden
  - Cardiologicum Dresden und Pirna - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Kreutzmann, Dresden
  - Herzzentrum Dresden GmbH Universitaetsklinik, Dresden
  - Uniklinik TU Dresden - Herzzentrum Dresden GmbH, Dresden
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - MVZ CCB Frankfurt Und Main-Taunus GbR, Frankfurt
  - Nephrologie Universitätsklinikum Frankfurt, Frankfurt
  - Uniklinik FFM - Nephrologie, Frankfurt
  - Studienzentrum ClinPhenomics, Frankfurt
  - Nierenzentrum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle - Innere Medizin II, Halle
  - St. Josefskrankenhaus Heidelberg - Diabeteszentrum, Heidelberg
  - Universitätsklinikum des Saarlandes - Innere Med. III, Homburg
  - Universitätsklinikum des Saarlandes - Innere Med. IV, Homburg Saar
  - Uniklinik Jena - Kardiologie, Jena
  - University Hospital Jena KöR, Jena
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Marienhaus Klinikum Mainz GmbH - Innere Medizin I, Mainz
  - Universitätsmedizin Mainz, Kardiologie I, Studienzentrum, Mainz
  - zero PRAXEN Mannheim-Schwetzingerstadt, Mannheim
  - Praxis Reichelsheim, Reichelsheim
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
  - Kahrmann, Witten
- Greece (30):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - University Hospital of Athens ATTIKON, Haidari-Athens, Attica
  - Alexandroupoli University General Hospital, Alexandroupoli
  - "Laiko" General Hospital of Athens, Athens
  - Hippokration Hospital, Athens
  - Thoracic General Hospital Of Athens I Sotiria - Cardiology Department, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - General Hospital of Chios "Skilitsio" - Cardiology Clinic, Chios
  - General Hospital of Chios "Skilitsio", Chios
  - Periphery University Hospital of Heraklion, Heraklion
  - University General Hospital Of Heraklion, Heraklion
  - University General Hospital of Ioannina,Internal Medicine, Ioannina
  - Kat Attica General Hospital - Cardiology Clinic, Kifissia
  - KAT General Hospital of Attica, Kifissia
  - General Hospital of Lamia, Lamia
  - Univ Gen Hospital Larisa, Cardiology Medicine Clinic, Larissa
  - Iatriko Athinon (Athens Medical Canter), Pylea, Thessaloniki
  - General University Hospital of Patras,Nephrology clinic, Rio, Patra
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - "AHEPA" University Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
  - General Hospital of Thessaloniki 'Ippokrateio' Dialysis Unit, Thessaloniki
  - General Hospital of Thessaloniki 'Agios Pavlos' - Nephrology Clinic, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - Iatriko Athinon (Athens Medical Canter), Thessaloniki
  - Gen Hospital of Thessaloniki G.Papanikolaou,Cardiology Dpt, Thessaloniki
- Hungary (9):
  - Dr. Lakatos Ferenc Kardiológus ,Belgyógyász Magán szakrendelés, Békéscsaba, Bekes County
  - Selye János Kórház, Komárom, Komárom-Esztergom
  - Léda Platán Magánklinika, Zalaegerszeg, Zala County
  - EURÉKA-CENTER Orvosi és Szolgáltató Betéti Társaság, Baja
  - Tagore Medical Center, Balatonfüred
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Jahn Ferenc Dél-pesti Kórház és Rendelőintézet, Budapest
  - DE KK Kardiológiai és Szívsebészeti klinika, Debrecen
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged
- India (49):
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - Vedanta Hospitals, Guntur, Andhra Pradesh
  - NIZAM'S Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Sunrise Hospital, Vijayawada, Andhra Pradesh
  - Apollo CHSF Heart Institute, Ahmedabad, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - Unicare heart institute and research centre, Surat, Gujarat
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - Manipal Hospital, Old Airport Road, Bengaluru, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bengaluru, Karnataka
  - Omega Hospital (P) Limited, Mangalore, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Manipal, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Karnataka
  - KLES & Prabhakar Kore Hospital and Research Centre, Belagavi, Karnatka
  - Lisie Hospital, Kochi, Kerala
  - Calicut Medical College, Kozhikode, Kerala
  - Government Medical College Trivandrum, Trivandrum, Kerala
  - Kamalnayan Bajaj Hospital, Aurangabad, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Government Medical College and Super Speciality Hospital, Nagpur, Nagpur, Maharashtra
  - Arneja Heart & Multispeciality Hospital, Nagpur, Maharashtra
  - Shri Krishna Hrudayalaya & Critical Care Centre, Nagpur, Maharashtra
  - Chopda Medicare and Research Centre Pvt. Ltd., Nashik, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - B J Goverment Medical College and Sassoon General Hospital, Pune, Maharashtra
  - Grant Medical Foundation, Pune, Maharashtra
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - Fortis Escorts Heart Institute, New Delhi, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Center, New Delhi, National Capital Territory of Delhi
  - VMMC & Safdarjung Hospital, New Dehli, New Delhi
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Apollo Hospitals Education & Research Foundation, Chennai, Tamil Nadu
  - Osmania General Hospital_Hyderabad, Hyderabad, Telangana
  - Osmania General Hospital, Hyderabad, Telangana
  - Guru Nanak CARE Hospitals, Hyderabad, Telangana
  - Apollo Hospital Jubilee Hills, Hyderabad, Hyderabad, Telangana
  - Osmania General Hospital, Hyderbad, Telangana
  - Gandhi Memorial Hospital- King George's Medical University, Lucknow, Uttar Pradesh
  - Medanta Lucknow Hospital, Lucknow, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, Chandigarh
  - Eternal Heart Care Centre, Jaipur
  - G B Pant Institute of Postgraduate Medical Education and Res, New Delhi
  - Lok Nayak Hospital, New Delhi
  - Max Super Speciality Hospital, Saket, New Delhi
  - Max Super Speciality Hospital_New Delhi, New Delhi
  - Fortis Escort Health Institute, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Lakshmi Hospital, Palakkad
- Israel (7):
  - Wolfson MC - Diabetes Clinic, Holon
  - Hadassah Ein Karam MC - Cardio Department, Jerusalem
  - Western Galilee MC - Cardiology Department, Nahariya
  - Rabin MC Beilinson - Cardiology department, Petah Tikva
  - Kaplan MC - Nephrology unit, Rehovot
  - Sourasky MC - Cardio Vascular Research Center, Tel Aviv
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
- Italy (24):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - A.O.U. Ferrara, Sant'Anna, Cona (Ferrara), Fe
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - Policlinico Umberto I Seconda Clinica Medica, Roma, RM
  - West Vicenza General Hospital, Arzignano (VI)
  - Policlinico S. Orsola - Malpighi, Bologna
  - AO Cannizzaro, Catania
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti Scalo
  - AOU Careggi Firenze, Florence
  - IRCCS Azienda Ospedaliero Universitaria San Martino - IST, Genova
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele S.r.l. - Unità Clinica Riabilitazione Specialistica Cardiologica, Milan
  - Centro Cardiologico Monzino, Milan
  - ASST degli Spedali Civili di Brescia-Presidio Ospedaliero di Montichiari, Montichiari
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - AOUP Giaccone Palermo, Palermo
  - ARNAS Ospedali Civico Di Cristina Benfratelli - Presidio Ospedaliero "Civio e Benfratelli", Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AOU Pisana Cisanello, Pisa
  - Policlinico Tor Vergata, Roma
  - Policlinico A. Gemelli IRCCS, Roma
  - AOU S. Andrea, Rome
  - Azienda Sanitaria Univ Giuliano Isontina, Trieste
  - AOUI Verona, Verona
- Japan (86):
  - Uwajima City Hospital_ Cardiology, Uwajima-shi, Ehime
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Seino Internal Medicine Clinic, Koriyama-shi, Fukushima, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Miyazaki Medical Association Hospital_Cardiology, Miyazaki, Miyazaki
  - NIPPON MEDICAL SCHOOL HOSPITAL_Cardiovascular medicine, Bunkyo-ku, Tokyo
  - The Univ. of Tokyo Hp., Dept. of Cardiovascular Medicine, Bunkyo-ku, Tokyo
  - Akaicho Clinic, Chiba-shi, Chiba
  - Fukuokaken Saiseikai Futsukaichi Hospital_Cardiovascular Medicine, Chikushino-shi, Fukuoka
  - University of Yamanashi Hospital_Cardiology, Chuo-city, Yamanashi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka-shi, Fukuoka
  - Fukuoka University Hospital_Cardiology, Fukuoka-shi, Fukuoka
  - National Hospital Organization Hamada Medical Center, Hamada-shi, Shimane
  - JA Shizuoka Kohseiren Enshu Hospital_ Cardiology, Hamamatsu-shi, Shizuoka
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - National Hospital Organization Mito Medical Center_Cardiovascular medicine, Ibaraki
  - Nishiyamado Keiwa Hospital_Internal Medicine, Ibaraki
  - Nishiyamado Keiwa Hospital, Ibaraki
  - Kishiwada Tokushukai Hospital_Cardiology, Kishiwada, Osaka
  - North Alps Medical Center Azumi Hospital_Cardiology, Kita-azumi-gun, Nagano
  - Steel Memorial Yawata Hospital_Cardiology, Kitakyushu-shi, Fukuoka
  - Kokura Memorial Hospital_Cardiology, Kitakyushu-shi,Fukuoka
  - National Hospital Organization Fukuokahigashi Medical Center, Koga-shi, Fukuoka
  - Kumamoto University Hospital, Cardiovascular Medicine, Kumamoto-shi, Kumamoto
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - Kyoto Okamoto Memorial Hospital_Cardiology, Kusegun, Kyoto
  - Kyoto Okamoto Memorial Hospital, Kusegun, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto-shi, Kyoto
  - National Hospital Organization Kyoto Medical Center_Cardiology, Kyoto-shi, Kyoto
  - Ijinkai Takeda General Hospital, Cardiovascular Medicine, Kyoto-shi,Kyoto
  - Maebashi Red Cross Hospital_Cardiology, Maebashi-shi, Gunma
  - Maebashi Red Cross Hospital, Maebashi-shi, Gunma
  - Matsubara Tokushukai Hospital_Neurosurgery, Matsubara-shi, Osaka
  - Chiba-Nishi General Hospital, Cardiology, Matsudo-shi
  - Shinshu University Hospital_Matsumoto-shi, Nagano, Matsumoto-shi, Nagano
  - Mishuku Hospital_Meguro-ku, Tokyo, Meguro-ku, Tokyo
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Hayama Heart Center, Miura-gun, Kanagawa
  - Miyakonojo Medical Association Hospital_Cardiology, Miyakonojo-shi, Miyazaki
  - Miyakonojo Medical Association Hospital, Miyakonojo-shi, Miyazaki
  - Iwate Prefectural Central Hospital_Cardiology, Morioka-shi, Iwate
  - Iwate Prefectural Central Hospital, Morioka-shi, Iwate
  - Social Medical Corporation Kojunkai Daido Clinic, Nagoya-shi, Aichi
  - Nagoya University Hospital_Nagoya-shi, Aichi, Nagoya-shi, Aichi
  - Naha City Hospital_Cardiovascular Medicine, Naha-shi, Okinawa
  - Naha City Hospital, Naha-shi, Okinawa
  - Nara Prefecture General Medical Center, Nara-shi, Nara
  - Hyogo Prefectual Nishinomiya Hospital_Nephrology, Nishinomiya-shi, Hyogo
  - Oita Medical Center_Cardiology, Oita-shi, Oita
  - Kawasaki Medical School Hospital, Okayama
  - Omihachiman Community Medical Center_Omihachiman-shi, Siga, Omihachiman-shi, Siga
  - Saiseikai Suita Hospital_Cardiovascular Medicine, Osaka
  - Takatsuki Red Cross Hospital_Diabetes and Endocrine Div., Osaka
  - Takatsuki Red Cross Hospital, Osaka
  - Yao Tokushukai General Hospital_Cardiovascular division, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka-city, Osaka
  - Yodogawa Christian Hospital, Osaka-shi, Osaka
  - Osaka City General Hospital_Osaka-shi, Osaka, Osaka-shi, Osaka
  - Kitada Clinic, Osaka-shi, Osaka
  - Social Corporation Keigakukai Minami Osaka Hospital_Cardiology, Osaka-shi,Osaka
  - Ota Memorial Hospital, Ota-shi, Gunma
  - Kitasato University Hospital_Sagamihara-shi, Kanagawa, Sagamihara-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Sagamihara-shi, Kanagawa
  - Sanai Hospital_Cardiology, Saitama-shi, Saitama
  - Sanai Hospital, Saitama-shi, Saitama
  - Hanaoka Seishu Memorial Hosp._Cardiovascular Medicine, Sapporo-shi, Hokkaido
  - Tohoku University Hospital, Cardiovascular, Sendai-shi, Miyagi
  - Sendai Cardiovascular Center_Cardiology, Sendai-shi, Miyagi
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
  - Saiseikai Suita Hospital_Suita-shi, Osaka, Suita-shi, Osaka
  - Osaka Saiseikai Senri Hospital_Cardiology, Suita-shi, Osaka
  - Osaka Saiseikai Senri Hospital, Suita-shi, Osaka
  - National Hospital Organization Disaster Medical Center_Nephrology, Tachikawa-shi, Tokyo
  - Takamatsu Red Cross Hospital_Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Kagawa Prefectural Central Hospital, Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Minamino Cardiovascular Hospital_Cardiovascular medicine, Tokyo
  - Saiseikai tondabayashi Hospital, Tondabayashi-shi, Osaka
  - Tsukuba Medical Center Hospital_Department of Cardiology, Tsukuba-shi, Ibaraki
  - Japanese Red Cross Wakayama Medical Center_Diabetology and Endocrinology, Wakayama
  - National Hospital Organization Saitama Hospital, Wako-shi, Saitama
  - Saiseikai Yokohamashi Nanbu Hospital_Cardiology, Yokohama-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama-shi, Kanagawa
  - Sanyudo Hospital_Cardiology, Yonezawa-shi, Yamagata
  - Sanyudo Hospital, Yonezawa-shi, Yamagata
- Latvia (6):
  - Ari Med, Daugavpils
  - Daugavpils Regional Hospital, Daugavpils
  - Zemgales diabetes centre, Jelgava
  - P. Stradins Clinical University Hospital, Riga
  - Adoria, Riga
  - Riga East Clinical University Hospital - Clinic "Gailezers", Riga
- Lithuania (12):
  - Klinikiniai sprendimai, Alytus, Alytus
  - Lithuanian university of health sciences Clinical hospital, Kaunas
  - Kaunas City Polyclinic, Silainiu department, Kaunas
  - Klinikiniai sprendimai, Kaunas, Kaunas
  - JSC "Saules seimos medicinos centras", Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Kaunas City polyclinic Dainava Branch, Kaunas
  - Klaipeda university hospital, Klaipėda
  - Republican Panevezys Hospital, Panevezys
  - Pirmoji Viltis, Šiauliai
  - JSC Inlita Lazdynai CMC, Vilnius
  - JSC Inlita Santaros, Vilnius
- Malaysia (15):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Sultan Abdul Halim, Sungai Petani, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Universiti Sains Malaysia_Kota Bharu, Kelantan, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - Hospital Miri, Miri, Sarawak
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - National Heart Institute, Kuala Lumpur
  - Hospital Seberang Jaya, Pulau Pinang
  - Hospital Queen Elizabeth II, Sabak Bernam
  - Hospital Tuanku Jaafar, Seremban
- Mexico (14):
  - CINCAME, Tijuana, Estado de Baja California
  - Consultorio Privado Dr Gabriel Arturo Ramos, Guadalajara, Jalisco
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - Clínicos Asociados BOCM, S.C., Benito Juárez, Mexico City
  - Clínicos Asociados BOCM, S.C., Mexico City, México, D.F.
  - Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Unidad Biomedica Avanzada Monterrey, Monterrey, Nuevo León
  - Centro de atención e investigación cardiovascular del Potosí, San Luis Potosí City, San Luis Potosí
  - Hospital Angeles de Culiacan, Culiacán, Sinaloa
  - Centro para el Desarrollo de la Medicina y la Asistencia, Culiacán, Sinaloa
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
  - Centro de Estudios Clínicos de Querétaro S.C., Querétaro
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (12):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuis Groep Twente Almelo, Almelo
  - Academisch Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Amphia Ziekenhuis, Breda
  - St Jansdal, Harderwijk
  - Tergooi, locatie Hilversum, Hilversum
  - Leids Universitair Medisch Centrum, Leiden
  - Bravis Ziekenhuis, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - D & A Research B.V., Sneek
  - Zaans Medisch Centrum, Zaandam
- Poland (34):
  - Kardio Life - Tomasz Borkowski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Zdrowie S.C. Agnieszka I Donald Drozdz, Wroclaw, Lower Silesian Voivodeship
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin, Lublin Voivodeship
  - ETG Poniatowa, Poniatowa, Lublin Voivodeship
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku K. Kardio, Bialystok, Podlaskie Voivodeship
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - Aka-Med Centrum, Ruda Śląska, Silesian Voivodeship
  - Poradnia Aka-Med Centrum Sp. z o.o., Ruda Śląska, Silesian Voivodeship
  - Centrum Kliniczno Badawcze, Elblag
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni Im.Sw.Jana Pawla II, Grodzisk Mazowiecki
  - Specjalistyczna Praktyka Lekarska L. Bryniarski, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Praktyka Lekarska Mateusz Sidor, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - Centrum Terapii Wspolczesnej, Lodz
  - Salve Medica, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Specjalistyczna Praktyka Lekarska w Ogrodzieńcu, Ogrodzieniec
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan
  - Velocity Nova Sp. z o.o., Puławy
  - CENTRUM MEDYCZNE VITA Praktyka Kardiologiczna, Szczecin
  - Polsko - Amerykanskie Kliniki Serca X Oddzial Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji w Tychach, Tychy
  - NBR Polska Tomasz Klodawski, Warsaw
  - Narodowy Instytut Kardiologii Klin. Kard. i Ang., Warsaw
  - Narodowy Instytut Kardiologii Klin. Kard. i Transp., Warsaw
  - Szpital Powiatowy Im. Hrabiego Stanislawa Lubienskiego Samodzielny Publiczny Zakład Opieki Zdrowotnej W Wegrowie, Węgrów
  - Centrum Badan Klinicznych, Wroclaw
  - Velocity Zamość, Zamość
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
- Portugal (14):
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital de Santa Cruz, Carnaxide, Lisbon District
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Unidade Local De Saude De Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade Local De Saude Da Regiao De Aveiro E.P.E., Aveiro
  - Unidade de Local de Saúde de Braga, Braga
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Unidade Local De Saude de Tâmega e Sousa E.P.E., Guilhufe - Penafiel
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital São Francisco Xavier, Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - Unidade Local de Saúde da Arrábida, E.P.E., Setúbal
  - Unidade Local de Saúde do Alto Minho E.P.E. - Viana do Castelo, Viana do Castelo
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- Romania (31):
  - Institutul Clinic Fundeni, Bucharest, Bucharest
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Clinic of Diabetes Cluj, Cluj-Napoca, Cluj
  - Cabinet Medical de Cardiologie Dr. Calin Pop, Baia Mare
  - S.C. Centrul Medical Unirea S.R.L., Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - Spitalul Județean de Urgență Brăila, Brăila
  - Hightech Medical Services S.R.L., Bucharest
  - Spitalul Universitar de Urgență Elias, Bucharest
  - Lotus Med SRL, Bucharest
  - Centrul Medical Emerald, Bucharest
  - Donna Medplus S.R.L., Bucharest
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest
  - Davius Clinicmed Srl, Bucharest
  - Spitalul Clinic de Urgenta "Sf. Ioan" Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Mat Cord Biomedica S.R.L., Buzău
  - Spitalul Clinic Judetean De Urgenta Sfantul Apostol Andrei Constanta, Constanța
  - Neurocord Medical SRL, Craiova
  - Cardiomed SRL, Craiova
  - SC Diamed Obesity SRL, Galati
  - Institutul de Boli Cardiovasculare "Prof. Dr. George I.M. Georgescu", Iași
  - SC Consultmed SRL, Iași
  - SC Cardiomed SRL, Iași
  - Spitalul Clinic Judetean De Urgenta Bihor, Oradea
  - Bella Praxis S.R.L., Paşcani
  - Sc Sal Med Srl, Piteşti
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - CMI Dr. Cristian Podoleanu, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
  - Institutul de Boli Cardiovasculare Timisoara, Timișoara
- Russia (21):
  - Reg. State Budget Healthc. Inst. Regional Clinical Hospital, Barnaul
  - RBSHI "Altay Regional Cardiology Dispensary", Barnaul
  - Road Clinical Hospital at station Chelyabinsk, Chelyabinsk
  - Chita State Medical Academy, Chita
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - FSB EI "Kazan' State Medical University", Kazan'
  - SAI of Health "Interregional Clinic Diagnostic Center", Kazan'
  - Institute of Complex Problems of Cardio-Vascular Diseases, Kemerovo
  - National Medical Research Center of Cardiology, Moscow
  - Pirogov Russian National Research Medical University MoH, Moscow
  - Friendship University of Russia MCCH base, Moscow
  - LLC RC Medical, Novosibirsk
  - State Novosibirsk regional clinical hospital, Novosibirsk
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - SBIH Perm region "City Clinical Hospital #2 n.a. F.K. Gral", Perm
  - Republican Hospital n.a. V. A. Baranov, Petrozavodsk
  - Medical Research Institute LLC, Saint Petersburg
  - SPb BHI "City Pokrovskaya Hospital", Saint Petersburg
  - Regional Clinical cardiological dispensary n.a. Polyakov, Samara
  - City Hospital #4, Sochi, Sochi
  - Tomsk National Research Medical Center of the RAS, Tomsk
- Serbia (12):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Clinical centre of Serbia, Clinic for cardiology, Belgrade
  - Clinical Centre of Serbia, Emergency Centre, Department of Cardiology, Belgrade
  - Emergency Internal Medicine Clinic, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Institute for Cardiovascular Diseases ''Dedinje'', Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Institute for Cardiovascular Diseases of Vojvodina - Sremska Kamenica, Kamenitz
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
  - University Clinical Centre Nis, Clinic for Cardiology, Niš
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad
- Slovakia (17):
  - CARDIOCONSULT, s.r.o., Bratislava
  - I. Interna klinika LF UK a UNB, Bratislava
  - DIABEDA s.r.o., Bratislava
  - 1. Interna klinika SZU a UNB, Bratislava
  - Klinika kardiologie a angiologie LF SZU, Bratislava
  - CINRE s. r. o., Oddelenie akutnej kardiologie a koronarna JIS, Bratislava
  - Medical group Kosice s.r.o., Košice
  - VITAL, s.r.o., Levice
  - KARDIO 1, s.r.o., Kardiologicka ambulancia, Lučenec
  - Narodny Endokrinologicky a diabetologicky ustav, Ľubochňa
  - 1. interna klinika, Univerzitna nemocnica Martin, Martin
  - InterStom, s.r.o., Nitra
  - KARDIOMED NZ, s.r.o., Nové Zámky
  - Medical KG, s.r.o., Piešťany
  - Kardiologicka ambulancia, Považská Bystrica
  - FNsP J. A. Reimana Presov, Klinika kardiologie, Prešov
  - IMCORE, s.r.o., Prešov
- South Africa (24):
  - Excellentis Clinical Trial Consultants, George, Eastern Cape
  - Cardiology Research_Bloemfontein, Bloemfontein, Free State
  - IATROS International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - Dr Iftikhar Osman Ebrahim, Centurion, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Tickerdoc Research (Pty) LTD, Johannesburg, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - EMMED Clinical Research, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Mediclinic Medical Centre, Tongaat, KwaZulu-Natal
  - Helderberg Research Institute, Cape Town, Western Cape
  - Tread Research (Pty)Ltd, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Prof Rayner_Division of Nephrology, Cape Town, Western Cape
  - TASK Eden Clinical Research Centre, George, Western Cape
  - Dr Hendrik Snyman's Practice, Mossel Bay, Western Cape
  - Paarl Reserch Centre, Paarl, Western Cape
  - Paarl Research Centre, Paarl, Cape Town, Western Cape
  - Clinical Trials Network Helderberg, Somerset West, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
- South Korea (25):
  - Dong-A University Hospital, Busan
  - Dong-A University Medical Center, Busan
  - Pusan National University Hospital, Busan
  - Daegu Catholic Univ. Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Wonju Severance Christian Hospital, Gangwon-do
  - National Health Insurance Corporation Ilsan Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Hanyang University GURI Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kyunghee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - KangNam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (12):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Univ. Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Reina Sofia, Córdoba
  - Bellvitge Universitary Hospital, L' Hospitalet Del Llobregat
  - Hospital Virgen del Camino - Sanlúcar de Barrameda, Sanlúcar de Barrameda
  - Hospital Vithas Sevilla, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Virgen de las Montañas, Villamartín
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (7):
  - Karolinska Universitetssjukhuset, Huddinge, Huddinge, Stockholm County
  - Njurmedicin, Gothenburg
  - Clemenstorgets Hjärtmottagning, Lund
  - Forskningsmottagning Internmedicin (tidigare KFE), Malmo
  - Njursektionen Medicinkliniken Örebro University Hospital, Örebro
  - Karolinska Universitetssjukhuset Solna,FOU Tema Hjärta Kärl, Stockholm
  - Forskning njurmedicin Uppsala, Uppsala
- Taiwan (11):
  - HsinChu MacKay Memorial Hospital, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital-Department of Cardiology, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei Medical University Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
  - National Yang Ming Chiao Tung University Hospital Lanyang Campus, Yilan
- Thailand (21):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Thammasat University Hospital, Klong Luang, Pathumthani, Changwat Pathum Thani
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Mueang Chiang Mai
  - King Chulalongkorn Memorial Hospital, Bangkok, Patumwan
  - Phramongkutklao Hospital_Nephrology, Bangkok, Rajathewee
  - Ramathibodi Hospital, Bangkok, Thung Phayathai Subdistrict
  - Chulabhorn hospital_Cardiovascular, Bangkok
  - Cardio-Vajira, Bangkok
  - Vajira Hospital - Cardio, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Rihes - Research Institute for Health Sciences, Chiang Mai
  - RIHES-CMU_Research Institute for Health Sciences, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Thammasat Hospital, Pathum Thani
  - Songklanagarind Hospital, Songkhla
  - Sunpasitthiprasong Hospital_Pediatrics Department, Ubon Ratchathani
  - Sunpasitthiprasong Hospital, Ubon Ratchathani
- Turkey (Türkiye) (27):
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi Hastanesi- Nefroloji, Istanbul, Bakirkoy
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul, Bakirkoy
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Afyonkarahisar Sağlık Bilimleri Üniversitesi Sağlık Uygulama Ve Araştırma Merkezi- Kardiyoloji, Afyonkarahisar
  - Hacettepe Universitesi Tip Fakultesi Nefroloji Bilim Dali, Ankara
  - Hacettepe University Medical Faculty_Ankara, Ankara
  - Hacettepe Üniversitesi Hastanesi- Kardiyoloji, Ankara
  - Hacettepe Üniversitesi Hastanesi- Nefroloji, Ankara
  - Ankara Bilkent Şehir Hastanesi-Kardiyoloji, Ankara
  - Akdeniz Universitesi Hastanesi Nefroloji Bilim Dali, Antalya
  - Akdeniz Üniversitesi Hastanesi-Nefroloji, Antalya
  - Aydın Adnan Menderes Üniversitesi Hastanesi- Nefroloji, Aydin
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Eskisehir Osmangazi University-Cardio, Eskişehir
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Kardiyoloji, Eskişehir
  - İstanbul Üniversitesi-Cerrahpaşa Tıp Fakültesi Kardiyoloji Enstitüsü, Istanbul
  - Istanbul Florence Nightingale Hospital, Istanbul
  - Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi EAH- Kardiyoloji, Istanbul
  - Ege Üniversitesi Hastanesi- Kardiyoloji, Izmir
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi-Kardiyoloji, Izmir
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş
  - Erciyes University Medial Faculty, Kayseri
  - Erciyes Üniversitesi Hastanesi- Nefroloji, Kayseri
  - Kocaeli University Nephrology Department, Kocaeli
  - Kocaeli Üniversitesi Araştıma ve Uygulama Hastanesi - Nefroloji, Kocaeli
  - Mersin Üniversitesi Hastanesi- Kardiyoloji, Mersin
  - Muğla Eğitim ve Araştırma Hastanesi, Muğla
- Ukraine (23):
  - Chernivtsi Emergency Hospital - Therapeutic Department No.1, Chernivtsi
  - Reg Clin Hospital of Emergency Care, Bukovinian Medical Univ, Chernivtsi
  - Сlinical treatment and diagnostic centre 'Simedgroup', Ivano-Frankivsk
  - City Clinical Hospital #27 (Kharkiv) - Intensive care department, Kharkiv
  - Institute of Therapy named after L.T.Malaya - Department of Prevention and Treatment of Kidney Diseases in Comorbid Conditions, Kharkiv
  - NI of Therapy na LT Malaya of NAMSU - Chr. Non-Communicable, Kharkiv
  - City Clinical Hospital #8 (Kharkiv) - Dept of Arterial and Ven Thrombosis, Kharkiv
  - Municipal Non-Profit Institution "City Clinical Hospital #8", Kharkiv
  - Medical Centre "OkClinic +" - inpatient department, Kyiv
  - Kyiv City Clinical Hospital of Emergency Care - Infarction department, Kyiv
  - Kyiv City Clinical Hospital of Emergency Care - Infarction, Kyiv
  - "Medbud-Clinic" LLC - medical and preventive unit, Kyiv
  - Medbud-Clinic LLC, Kyiv
  - Clinical Hosp on the railway line №2 branch PHC JSC Ukrzaliz, Kyiv
  - Kyiv Railway Clinical Hospital #2 - day care department, Kyiv
  - M.D.Strazheska Institute of Cardiology of NAMSU - Intensive care and resuscitation department, Kyiv
  - M.D.Strazheska Institute of Cardiology of NAMSU - Department of non-coronary heart diseases, Kyiv
  - Medical Center 'Consilium Medical' - clinical consultation department, Kyiv
  - Kyiv Regional Clinical Hospital - Consultative medical department, Kyiv
  - "Center of Family Medicine Plus" LLC - Outpatient department, Kyiv
  - City Clinical Hospital #10 (Zaporizhia) - Therapeutics department, Zaporizhia
  - University Clinic of Zaporizhia State Medical and Pharm University - Cardiology department, Zaporizhzhia
  - Central City Hospital #1 - Scientific-Research centre, Zhytomyr
- United Kingdom (35):
  - Ashfields Primary Care Centre, Sandbach, Cheshire
  - Royal Bournemouth Hospital - Cardiology, Bournemouth, Dorset
  - Dorset County Hospital, Dorchester, Dorset
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Pickering Medical Practice, Pickering, North Yorkshire
  - Lakeside Healthcare Research & Innovation Unit, Corby, Northamptonshire
  - Crouch Oak Family Practice, Addlestone, Surrey
  - St. Richards Hospital_Cardiology, Chichester, West Sussex
  - Barnet Hospital - Cardiology Department, Barnet
  - Sandwell General Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital - Cambridge Dialysis Centre, Cambridge
  - The Adam Practice, Dorset
  - Carmel Medical Practice, Durham
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Wycombe General Hospital, High Wycombe
  - Cardiology, Leicester
  - Leicester General Hospital, Leicester
  - Lincoln County Hospital, Lincoln
  - Liverpool Heart & Chest Hospital, Liverpool
  - Aintree University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - William Harvey Clinical Research Centre, London
  - Kings College Hospital, London
  - Freeman Hospital, Newcastle, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford
  - Panthera Biopartners Preston, Preston
  - Sherbourne Medical Centre, Royal Leamington Spa
  - Lister Hospital, Stevenage
  - University of North Tees Hospital, Stockton-on-Tees
  - Musgrove Park Hospital, Taunton
  - Cardiology Department, Torquay
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Byambaa E, Roshanravan B, Berglund L. Lipoprotein(a) and CKD: Insights into New Therapeutic Opportunities. Clin J Am Soc Nephrol. 2025 Dec 2. doi: 10.2215/CJN.0000000968. Online ahead of print. PMID 41329869
- [Derived] Mohammadnia N, van Broekhoven A, Bax WA, Eikelboom JW, Mosterd A, Fiolet ATL, Tijssen JGP, Thompson PL, de Kleijn DPV, Tsimikas S, Cornel JH, Yeang C, El Messaoudi S. Interleukin-6 modifies Lipoprotein(a) and oxidized phospholipids associated cardiovascular disease risk in a secondary prevention cohort. Atherosclerosis. 2025 Jun;405:119211. doi: 10.1016/j.atherosclerosis.2025.119211. Epub 2025 Apr 26. PMID 40318255